CLINICAL TRIAL: NCT00519597
Title: Randomized Intervention With CPAP in Coronary Artery Disease and Sleep Apnea - RICCADSA Trial
Brief Title: Continuous Positive Airway Pressure (CPAP) Treatment in Coronary Artery Disease and Sleep Apnea
Acronym: RICCADSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Skaraborg Hospital (Other Government)
Collaborators: The Swedish Research Council (Other Government); Swedish Heart Lung Foundation (Other); Heart Foundation of Karnsjukhuset Sweden (Unknown); ResMed Foundation (Other)
Responsible Party: Principal Investigator, Yuksel Peker, MD, PhD, Associate Professor, Skaraborg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGSKAS-4731
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Coronary Artery Disease; Obstructive Sleep Apnea
Keywords: Coronary Artery Disease; Sleep Apnea; CPAP; Revascularization; Mortality
MeSH Terms: conditions — Coronary Artery Disease; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- I (Experimental): Asymptomatic OSA (CPAP)
  Interventions: Device: ResMed S8 (Auto-CPAP)
- II (No Intervention): Asymptomatic OSA (no CPAP)
- III (Active Comparator): Symptomatic OSA (OSAS)
  Interventions: Device: ResMed S8 (Auto-CPAP)
- IV (No Intervention): Non-OSA

INTERVENTIONS:
Device: ResMed S8 (Auto-CPAP) — AutoCPAP during sleep
  Arms: I; III

SUMMARY:
Obstructive sleep apnea (OSA) worsens the prognosis in patients with coronary artery disease (CAD). Many of these subjects do not report daytime sleepiness, and therefore, are not considered for OSA treatment with continuous positive airway pressure (CPAP). There is lack of evidence regarding the impact of CPAP on the long-term prognosis of CAD patients with OSA. The Randomized Intervention with CPAP in CAD and OSA (RICCADSA) trial is designed to address if CPAP treatment reduces the combined rate of new revascularization, myocardial infarction, stroke and cardiovascular mortality over mean follow-up period of 3-years in CAD patients with OSA without daytime sleepiness.Secondary outcomes include cardiovascular biomarkers, cardiac function, maximal exercise capacity and quality of life at baseline, 3-month- and 1-year follow-up as well as polysomnographic findings and adherence to CPAP therapy.

DETAILED DESCRIPTION:
Rationale: OSA is a common condition in CAD with a poor prognosis.Many of these subjects do not report daytime sleepiness, and therefore, are not considered for OSA treatment with CPAP. There is lack of evidence regarding the impact of CPAP on the long-term prognosis of CAD patients with OSA.

Objective: The RICCADSA trial is designed to address if CPAP treatment reduces the combined rate of new revascularization, myocardial infarction, stroke and cardiovascular mortality over a mean follow-up period of 3-years in CAD patients with OSA (Apnea-Hypopnea-Index [AHI]>=15 per h) without daytime sleepiness (Epworth Sleepiness Scale [ESS]<10). Secondary outcomes include cardiovascular biomarkers, cardiac function, maximal exercise capacity and quality of life at baseline, 3-month- and 1-year follow-up as well as polysomnographic findings and adherence to CPAP therapy.

Patients and Methods: A sample of 511 CAD patients (122 non-sleepy OSA patients randomized to CPAP, 122 to non-CPAP; 155 sleepy OSA patients [ESS>=10] on CPAP, and 112 CAD patients without OSA [AHI <5 per h]) were included. The trial has 80% power to detect a risk reduction from an assumed composite end-point rate of 25% to 12% for the primary outcome at intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with angiographically-verified CAD who have newly undergone PCI or CABG treatment
* Written, informed study consent
* OSA (AHI>=15 per hour) or non-OSA (AHI<5 per hour) diagnosis on the unattended sleep recording at home

Exclusion Criteria:

* Patients with already treated OSAS
* Patients presenting mainly central apneas (Cheynes-Stokes breathing)
* Patients with borderline OSA (AHI <15 and >=5 per hour) upon the unattended sleep recording at home

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2005-12; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The combined rate of cardiovascular mortality, stroke, myocardial infarction and the need for a new revascularization. | Three years

SECONDARY OUTCOMES:
Cardiovascular biomarkers, left ventricular function, maximal exercise capacity, quality of life, anxiety and depression state. | Three months and one year, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Yüksel Peker, Ass. Prof., Study Chair — Göteborg University
Locations (1):
- Skaraborg Hospital, Skövde, Sweden

REFERENCES:
- [Result] Baniak LM, Chasens ER, Luyster FS, Strollo PJ Jr, Thunstrom E, Peker Y. Obstructive sleep apnea and self-reported functional impairment in revascularized patients with coronary artery disease in the RICCADSA trial. Sleep Breath. 2018 Dec;22(4):1169-1177. doi: 10.1007/s11325-018-1733-4. Epub 2018 Oct 15. PMID 30324547
- [Result] Balcan B, Thunstrom E, Strollo PJ Jr, Peker Y. Continuous Positive Airway Pressure Treatment and Depression in Adults with Coronary Artery Disease and Nonsleepy Obstructive Sleep Apnea. A Secondary Analysis of the RICCADSA Trial. Ann Am Thorac Soc. 2019 Jan;16(1):62-70. doi: 10.1513/AnnalsATS.201803-174OC. PMID 30130421
- [Result] Luyster FS, Strollo PJ Jr, Thunstrom E, Peker Y. Long-term use of continuous positive airway pressure therapy in coronary artery disease patients with nonsleepy obstructive sleep apnea. Clin Cardiol. 2017 Dec;40(12):1297-1302. doi: 10.1002/clc.22827. Epub 2017 Dec 14. PMID 29243273
- [Result] Peker Y, Thunstrom E, Glantz H, Wegscheider K, Eulenburg C. Outcomes in coronary artery disease patients with sleepy obstructive sleep apnoea on CPAP. Eur Respir J. 2017 Dec 7;50(6):1700749. doi: 10.1183/13993003.00749-2017. Print 2017 Dec. PMID 29217597
- [Result] Thunstrom E, Glantz H, Yucel-Lindberg T, Lindberg K, Saygin M, Peker Y. CPAP Does Not Reduce Inflammatory Biomarkers in Patients With Coronary Artery Disease and Nonsleepy Obstructive Sleep Apnea: A Randomized Controlled Trial. Sleep. 2017 Nov 1;40(11). doi: 10.1093/sleep/zsx157. PMID 29029237
- [Result] Glantz H, Johansson MC, Thunstrom E, Guron CW, Uzel H, Saygin M, Herlitz J, Peker Y. Effect of CPAP on diastolic function in coronary artery disease patients with nonsleepy obstructive sleep apnea: A randomized controlled trial. Int J Cardiol. 2017 Aug 15;241:12-18. doi: 10.1016/j.ijcard.2017.03.100. Epub 2017 Mar 25. PMID 28408103
- [Result] Peker Y, Wegscheider K, Eulenburg C. Reply: Effect of Continuous Positive Airway Pressure Therapy on Cardiovascular Outcomes: Risk Assessment. Am J Respir Crit Care Med. 2017 Sep 1;196(5):662-663. doi: 10.1164/rccm.201702-0420LE. No abstract available. PMID 28296427
- [Result] Peker Y, Glantz H, Eulenburg C, Wegscheider K, Herlitz J, Thunstrom E. Effect of Positive Airway Pressure on Cardiovascular Outcomes in Coronary Artery Disease Patients with Nonsleepy Obstructive Sleep Apnea. The RICCADSA Randomized Controlled Trial. Am J Respir Crit Care Med. 2016 Sep 1;194(5):613-20. doi: 10.1164/rccm.201601-0088OC. PMID 26914592
- [Result] Glantz H, Thunstrom E, Johansson MC, Wallentin Guron C, Uzel H, Ejdeback J, Nasic S, Peker Y. Obstructive sleep apnea is independently associated with worse diastolic function in coronary artery disease. Sleep Med. 2015 Jan;16(1):160-7. doi: 10.1016/j.sleep.2014.08.018. Epub 2014 Nov 18. PMID 25547036
- [Result] Thunstrom E, Glantz H, Fu M, Yucel-Lindberg T, Petzold M, Lindberg K, Peker Y. Increased inflammatory activity in nonobese patients with coronary artery disease and obstructive sleep apnea. Sleep. 2015 Mar 1;38(3):463-71. doi: 10.5665/sleep.4510. PMID 25325463
- [Result] Glantz H, Thunstrom E, Herlitz J, Cederin B, Nasic S, Ejdeback J, Peker Y. Occurrence and predictors of obstructive sleep apnea in a revascularized coronary artery disease cohort. Ann Am Thorac Soc. 2013 Aug;10(4):350-6. doi: 10.1513/AnnalsATS.201211-106OC. PMID 23952854
- [Result] Peker Y, Glantz H, Thunstrom E, Kallryd A, Herlitz J, Ejdeback J. Rationale and design of the Randomized Intervention with CPAP in Coronary Artery Disease and Sleep Apnoea--RICCADSA trial. Scand Cardiovasc J. 2009 Feb;43(1):24-31. doi: 10.1080/14017430802276106. PMID 18663661
- [Derived] Peker Y, Celik Y, Zinchuk A, Sands SA, Redline S, Azarbarzin A. Association of Hypoxic Burden With Cardiovascular Events: A Risk Stratification Analysis of the Randomized Intervention With CPAP in Coronary Artery Disease and Sleep Apnea Cohort. Chest. 2025 Dec;168(6):1481-1493. doi: 10.1016/j.chest.2025.07.4081. Epub 2025 Aug 14. PMID 40818776
- [Derived] Balcan B, Celik Y, Strollo PJ, Peker Y. Characteristics of short REM sleepers and long-term CPAP use in the RICCADSA cohort. Sleep Med. 2025 Sep;133:106647. doi: 10.1016/j.sleep.2025.106647. Epub 2025 Jun 19. PMID 40544785
- [Derived] Sanchez-de-la-Torre M, Gracia-Lavedan E, Benitez ID, Sanchez-de-la-Torre A, Moncusi-Moix A, Torres G, Loffler K, Woodman R, Adams R, Labarca G, Dreyse J, Eulenburg C, Thunstrom E, Glantz H, Peker Y, Anderson C, McEvoy D, Barbe F. Adherence to CPAP Treatment and the Risk of Recurrent Cardiovascular Events: A Meta-Analysis. JAMA. 2023 Oct 3;330(13):1255-1265. doi: 10.1001/jama.2023.17465. PMID 37787793
- [Derived] Eulenburg C, Celik Y, Redline S, Thunstrom E, Glantz H, Strollo PJ Jr, Peker Y. Cardiovascular Outcomes in Adults with Coronary Artery Disease and Obstructive Sleep Apnea with versus without Excessive Daytime Sleepiness in the RICCADSA Cinical Trial. Ann Am Thorac Soc. 2023 Jul;20(7):1048-1056. doi: 10.1513/AnnalsATS.202208-676OC. PMID 36800433
- [Derived] Peker Y, Holtstrand-Hjalm H, Celik Y, Glantz H, Thunstrom E. Postoperative Atrial Fibrillation in Adults with Obstructive Sleep Apnea Undergoing Coronary Artery Bypass Grafting in the RICCADSA Cohort. J Clin Med. 2022 Apr 27;11(9):2459. doi: 10.3390/jcm11092459. PMID 35566586
- [Derived] Celik Y, Balcan B, Peker Y. CPAP Intervention as an Add-On Treatment to Lipid-Lowering Medication in Coronary Artery Disease Patients with Obstructive Sleep Apnea in the RICCADSA Trial. J Clin Med. 2022 Jan 5;11(1):273. doi: 10.3390/jcm11010273. PMID 35012012
- [Derived] Reynor A, McArdle N, Shenoy B, Dhaliwal SS, Rea SC, Walsh J, Eastwood PR, Maddison K, Hillman DR, Ling I, Keenan BT, Maislin G, Magalang U, Pack AI, Mazzotti DR, Lee CH, Singh B. Continuous positive airway pressure and adverse cardiovascular events in obstructive sleep apnea: are participants of randomized trials representative of sleep clinic patients? Sleep. 2022 Apr 11;45(4):zsab264. doi: 10.1093/sleep/zsab264. PMID 34739082
- [Derived] Behboudi A, Thelander T, Yazici D, Celik Y, Yucel-Lindberg T, Thunstrom E, Peker Y. Association of TNF-alpha (-308G/A) Gene Polymorphism with Circulating TNF-alpha Levels and Excessive Daytime Sleepiness in Adults with Coronary Artery Disease and Concomitant Obstructive Sleep Apnea. J Clin Med. 2021 Jul 31;10(15):3413. doi: 10.3390/jcm10153413. PMID 34362196
- [Derived] Zinchuk AV, Chu JH, Liang J, Celik Y, Op de Beeck S, Redeker NS, Wellman A, Yaggi HK, Peker Y, Sands SA. Physiological Traits and Adherence to Sleep Apnea Therapy in Individuals with Coronary Artery Disease. Am J Respir Crit Care Med. 2021 Sep 15;204(6):703-712. doi: 10.1164/rccm.202101-0055OC. PMID 34156917
- [Derived] Celik Y, Thunstrom E, Strollo PJ Jr, Peker Y. Continuous positive airway pressure treatment and anxiety in adults with coronary artery disease and nonsleepy obstructive sleep apnea in the RICCADSA trial. Sleep Med. 2021 Jan;77:96-103. doi: 10.1016/j.sleep.2020.11.034. Epub 2020 Dec 4. PMID 33341644
- [Derived] Peker Y, Thunstrom E, Glantz H, Eulenburg C. Effect of Obstructive Sleep Apnea and CPAP Treatment on Cardiovascular Outcomes in Acute Coronary Syndrome in the RICCADSA Trial. J Clin Med. 2020 Dec 15;9(12):4051. doi: 10.3390/jcm9124051. PMID 33333899
- [Derived] Wallstrom S, Balcan B, Thunstrom E, Wolf A, Peker Y. CPAP and Health-Related Quality of Life in Adults With Coronary Artery Disease and Nonsleepy Obstructive Sleep Apnea in the RICCADSA Trial. J Clin Sleep Med. 2019 Sep 15;15(9):1311-1320. doi: 10.5664/jcsm.7926. PMID 31538602